CLINICAL TRIAL: NCT04919356
Title: G2019S LRRK2 Parkinson's Disease: Increasing Awareness and Genetic Testing Program
Brief Title: Parkinson's Disease G2019S LRRK2 Genetic Testing Program
Status: Terminated | Type: Observational
Why Stopped: Sponsor stopped the study
Sponsor: Escape Bio, Inc. (Industry)
Collaborators: Engage Health Inc. (Industry); Sano (Other)
Responsible Party: Sponsor
Other Study IDs: G2019S-001
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-08

CONDITIONS: Parkinson's Disease
Keywords: G2019S LRRK2 Mutation; Young Onset; Genetic; Ashkenazi Jewish Descent; North African Berber
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Data generation using next-generation sequencing (NGS) of human exons

INTERVENTIONS:
Genetic: G2019S LRRK2 — No cost genetic testing for G2019S LRRK2

SUMMARY:
Increase awareness of the G2019S LRRK2 mutation in Parkinson's and no cost genetic testing program.

DETAILED DESCRIPTION:
This program is intended to increase awareness of genetic Parkinson's, in particular the G2019S LRRK2 mutation, and provide no cost genetic testing to determine if they carry the G2019S LRRK2 mutation.

ELIGIBILITY:
Participants include those with a clinical diagnosis of Parkinson's, in particular those who have a first- or second-degree relative with Parkinson's, or who have young onset Parkinson's (age less than 50 at diagnosis) or are of Ashkenazi Jewish or North African Berber descent, or have a relative with a known genetic mutation in the LRRK2 gene, or who have a genetic mutation in the LRRK2 gene.

Inclusion Criteria:

Participant eligible for enrollment in the program must meet all of the following criteria:

1. Participant must be a person diagnosed with Parkinson's disease who is 18 years or older.
2. Participant is under the care of a physician for their Parkinson's disease.
3. Participant is able to read, write and understand English, and reside in a country where the shipment of biological samples is allowed.
4. Participant is able to grant informed consent.
5. In the case of participants, willing to participate in a free genetic testing program to determine if they carry the G2019S LRRK2 mutation.
6. Willing to be notified of eligibility for clinical studies (if appropriate).
7. Particpants who already believe they have tested positive for the mutation will be allowed to be retested through this program and be notified of potential eligibility for studies.

Exclusion Criteria:

1. Inability to meet any of the inclusion criteria.
2. Participant has received on of the following advanced treatments to manage their Parkinson's: gene therapy, deep brain stimulation (DBS), injections into the brain, continuous infusion of medication into their stomach/intestines with a pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A clinical diagnosis of Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Identify Parkinson's patients with the G2019S mutation in their LRRK2 gene | 2 years
  To identify Parkinson's patients with the G2019S mutation in their LRRK2 gene through whole exome sequencing in order to support the development of an oral precision medicine.

SECONDARY OUTCOMES:
Understand the proportion of Parkinson's patients who have a G2019S LRRK2 mutation | 2 years
  To obtain information about the proportion of Parkinson's patients who have a G2019S LRRK2 mutation.
Increase awareness of the importance of genetic testing in Parkinson's disease | 2 years
  To increase healthcare provider and patient awareness of the importance of genetic testing in Parkinson's disease in order to be aware of potential eligibility for clinical studies of genetic targeted medicines.
Increase interest of healthcare providers and patients participation in clinical trials | 2 years
  To engage healthcare providers and patients' interest in participation in upcoming clinical studies.

CONTACTS AND LOCATIONS:
Overall Officials: Carrolee Barlow, MD, PhD, Study Chair — ESCAPE Bio
Locations (1):
- Eurofins Genomic LLC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bright JM, Carlisle HJ, Toda AMA, Murphy M, Molitor TP, Wren P, Andruska KM, Liu E, Barlow C. Differential Inhibition of LRRK2 in Parkinson's Disease Patient Blood by a G2019S Selective LRRK2 Inhibitor. Mov Disord. 2021 Jun;36(6):1362-1371. doi: 10.1002/mds.28490. Epub 2021 Feb 11. PMID 33836114